CLINICAL TRIAL: NCT00659737
Title: A Randomized, Double-blind Comparison of Oral Aprepitant Alone Versus Oral Aprepitant and Transdermal Scopolamine for Preventing Postoperative Nausea and Vomiting
Brief Title: Comparison of Oral Aprepitant and Transdermal Scopolamine for Preventing Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University College of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20071433
Record Dates: First submitted 2008-04-08; First posted 2008-04-16 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2013-09

CONDITIONS: Nausea; Vomiting
Keywords: Post-operative Nausea and Vomiting (PONV)
MeSH Terms: conditions — Nausea; Vomiting | interventions — Aprepitant; Scopolamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant (Placebo Comparator): Oral Aprepitant pill and placebo transdermal patch at least 1 hour prior to surgical procedure.
  Emend (Aprepitant) + Placebo
  Interventions: Drug: Aprepitant
- Scopolamine (Active Comparator): Oral Aprepitant pill and Scopolamine transdermal patch at least 1 hour prior to surgical procedure.
  Interventions: Drug: Scopolamine

INTERVENTIONS:
Drug: Aprepitant — 40mg tablet
  Other Names: Emend (Aprepitant) + Placebo
  Arms: Aprepitant
Drug: Scopolamine — 1.5 mg patch delivering transdermally in vivo approx. 1.0mg over 3 days
  Other Names: Scopolamine + Emend (Aprepitant)
  Arms: Scopolamine

SUMMARY:
Recent evidence suggests multiple drug therapy is superior to single agents. The study compares the incidence of nausea, vomiting, need for rescue medication, prolonged PACU time, and unplanned hospital admission in patients with high risk for PONV treated with oral aprepitant with or without transdermal scopolamine preoperatively.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a serious problem complicating surgery. PONV has an overall incidence of 30% and a 70% incidence in high-risk patients. PONV yields unplanned hospital admission, pulmonary aspiration, esophageal rupture, electrolyte abnormalities, dehydration, and delayed discharge from the postanesthesia care unit (PACU). Additional use of resources costs the health care industry hundreds of millions of dollars annually. Patient satisfaction is greatly improved when PONV is prevented.4 PONV etiology is multifactorial and the treatment is multimodal.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be between 18 and 65 years of age.
* Patient's ASA (American Society of Anesthesiologist) class must be between 1 and 3.
* If patient is currently on oral contraceptive to prevent pregnancy, she must be willing to use a back up form of birth control for one month post study.
* Patient must have 1 FACTOR to qualify

  * Female Sex
  * History of PONV
  * Motion Sickness
  * Non-Smoker
  * Intended Use of Post Operative Opioids

Exclusion Criteria:

* Patients with a history of vomiting due to middle ear infection, nervous system disorder, or any other condition.
* The surgical procedure is less than 1 hour.
* The patient is pregnant or breast feeding.
* The patient has taken antiemetic medication in previous 24 hours.
* Patients with narrow-angle glaucoma.
* Allergy to belladonna alkaloids.
* Hypersensitivity to barbiturates.
* Patient taking any of the following medications:

  * Orap
  * Seldane
  * Hismanal
  * Propulsid
  * Phenytoin
  * Phenothiazines
  * Tricyclic Antidepressants
  * Meperidine
  * Tolbutamide
  * Aluminum and Magnesium Trisilicate-containing Antacids
  * Anti-Cholinergics
  * Coumadin
* Male patients with prostate hypertrophy.
* Patients with severe hepatic disease.
* Patients on Chemotherapy and taking Aprepitant.
* Patients with fever.
* Patients with sepsis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2008-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Horrow, MD, Study Director — Drexel University College of Medicine
Locations (1):
- Hahnemann University Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aprepitant and Placebo Transdermal Patch: Oral Aprepitant pill 40 mg tablet and placebo transdermal patch at least 1 hour prior to surgical procedure.
- Aprepitant and Scopolamine Transdermal Patch: Oral Aprepitant pill, 40 mg tablet and Scopolamine transdermal patch, 1.5 mg patch delivering transdermally in vivo approximately 1.0mg over 3 days, at least 1 hour prior to surgical procedure.
Period: Overall Study
Arm/Group | Aprepitant and Placebo Transdermal Patch | Aprepitant and Scopolamine Transdermal Patch
Started | 57 | 58
Completed | 57 | 58
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aprepitant and Placebo Transdermal Patch: Oral Aprepitant pill, 40 mg tablet and placebo transdermal patch at least 1 hour prior to surgical procedure.
- Total: Total of all reporting groups
Arm/Group | Aprepitant and Placebo Transdermal Patch | Aprepitant and Scopolamine Transdermal Patch | Total
Number analyzed (Participants) | 57 | 58 | 115
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.2 (11.27) | 46.3 (11.06) | 46.8 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 51 | 103
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Nausea and Vomiting
Time Frame: 0-24 hours
Measure: Number; unit: participants
Arm/Group | Aprepitant and Placebo Transdermal Patch | Aprepitant and Scopolamine Transdermal Patch
Number analyzed (Participants) | 57 | 58
participants | 28 | 34

ADVERSE EVENTS:
Time Frame: 0-24 hours
Groups:
- Aprepiatnt: Oral Aprepitant pill and placebo transdermal patch at least 1 hour prior to surgical procedure.
  Emend (Aprepitant) + Placebo: 40mg tablet
- Scopolamine: Oral Aprepitant pill and Scopolamine transdermal patch at least 1 hour prior to surgical procedure.
  Scopolamine + Emend (Aprepitant): 1.5 mg patch delivering transdermally in vivo approx. 1.0mg over 3 days
Arm/Group | Aprepiatnt | Scopolamine
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/58
Other Adverse Events (participants affected / at risk) | 29/57 | 34/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepiatnt (N=57) | Scopolamine (N=58)
Dry mouth (Gastrointestinal disorders) | 29 (29) | 34 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No